CLINICAL TRIAL: NCT03835572
Title: Evaluation of Circadian Health Educational Tool
Brief Title: CircaHealth Development and Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Quantum Foundation (Unknown)
Responsible Party: Principal Investigator, Dylan Petkus, Student Doctor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20180932
Record Dates: First submitted 2019-02-05; First posted 2019-02-08 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Health Behavior; Health Knowledge, Attitudes, Practice; Circadian Rhythm
Keywords: Circadian Rhythm; Education; Student burnout; Sleep Hygiene
MeSH Terms: conditions — Health Behavior; Behavior; Burnout, Psychological; Sleep Hygiene | interventions — Health

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to receive the online educational course or materials on sleep hygiene for six weeks.
Who Masked: Investigator
Masking Description: Participants will be assigned a study ID such that the investigators cannot determine the identify of the participants or which arm of the study each participant is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CircaHealth (Experimental): The CircaHealth group will receive access to an online educational module on circadian rhythms and health as their intervention. Every week for six weeks, these participants will receive a new module that contains videos, quizzes, behavioral modification checklists, and journal prompts.
  Interventions: Other: CircaHealth: a course on circadian rhythms and health
- Sleep hygiene materials (Active Comparator): The control group will receive publicly available materials about sleep hygiene from the National Sleep Foundation and/or the American Academy of Sleep Medicine every week for six weeks as their intervention.
  Interventions: Other: Sleep hygiene materials

INTERVENTIONS:
Other: CircaHealth: a course on circadian rhythms and health — Participants will receive videos, behavioral modification checklists, and quizzes every week for six weeks.
  Arms: CircaHealth
Other: Sleep hygiene materials — Participants in the control group will receive weekly materials from the National Sleep Foundation and American Academy of Sleep Medicine on sleep hygiene
  Arms: Sleep hygiene materials

SUMMARY:
This study evaluates the feasibility, acceptability, and efficacy of an online education course about circadian rhythms and health. Half of participants will be enrolled into the online course and the other half will receive materials on sleep hygiene as a control.

DETAILED DESCRIPTION:
This is a pilot randomized controlled study that aims to develop CircaHealth: an online course on practices, known as circadian hygiene, that promote circadian rhythm alignment and minimize circadian rhythm misalignment. The project also will determine the feasibility, acceptability, and preliminary effects of CircaHealth in improving circadian rhythm related measures in University of Miami Miller School of Medicine medical students.

The educational videos will be incorporated into a six-module online course which contains additional educational and behavior modification tools. Medical students (n = 40) will be recruited via email and randomized to receive CircaHealth or materials from the National Sleep Foundation and/or the American Academy of Sleep Medicine. Sleep, mood, and circadian hygiene knowledge, behaviors, and attitudes will be assessed at baseline and four weeks post intervention. Feasibility will be determined by CircaHealth module completion rates, and acceptability will be assessed via a self-report survey. Changes in sleep quality measures between groups will determine the preliminary efficacy of CircaHealth.

ELIGIBILITY:
Inclusion Criteria:

* Medical students, 1st through 4th year, at the University of Miami Miller School of Medicine willing to participate in surveys and the CircaHealth course.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-02-23 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
Participant completion rate of CircaHealth | Six weeks
  Determine how many participants completed all modules within CircaHealth. Participants status in the course will be assessed via survey weekly such that their completion of each module can be determined.
Participant qualitative feedback on CircaHealth | Six weeks
  Participants will be surveyed every week on what aspects of CircaHealth were helpful and what aspects of CircaHealth can be improved. This qualitative data will be analyzed to determine which aspects of CircaHealth positively and negatively impacted the educational value of the course.

SECONDARY OUTCOMES:
Change in Epworth Sleepiness Scale scores four weeks after the completion of CircaHealth | Ten weeks
  To determine if Epworth Sleepiness Scale scores improved four weeks after completion of the educational intervention in comparison to the control group.
Change in Pittsburgh Sleep Quality Index scores four weeks after the completion of CircaHealth | Ten weeks
  To determine if Pittsburgh Sleep Quality Index scores improved four weeks after completion of the educational intervention in comparison to the control group.
Change in Munich Chronotype scores four weeks after the completion of CircaHealth | Ten weeks
  To determine if Munich Chronotype scores improved four weeks after completion of the educational intervention in comparison to the control group.
Change in Circadian Health Scale scores four weeks after the completion of CircaHealth | Ten weeks
  To determine if Circadian Health Scale scores improved four weeks after completion of the educational intervention in comparison to the control group.
Change in Maslach General Survey for Students scores four weeks after the completion of CircaHealth | Ten weeks
  To determine if Maslach General Survey for Students scores improved four weeks after completion of the educational intervention in comparison to the control group.

OTHER OUTCOMES:
Association between Epworth Sleepiness Scale scores and Circadian Health Scale scores | Ten weeks
  To determine if Epworth Sleepiness Scale scores are associated with Circadian Health Scale scores
Association between Pittsburgh Sleep Quality Index scores and Circadian Health Scale scores | Ten weeks
  To determine if Pittsburgh Sleep Quality Index scores are associated with Circadian Health Scale scores
Association between Munich Chronotype scores and Circadian Health Scale scores | Ten weeks
  To determine if Munich Chronotype scores are associated with Circadian Health Scale scores
Association between Maslach General Survey for Students scores and Circadian Health Scale scores | Ten weeks
  To determine if Maslach General Survey for Students scores are associated with Circadian Health Scale scores

CONTACTS AND LOCATIONS:
Overall Officials: Tulay Koru-Sengal, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No